CLINICAL TRIAL: NCT06406439
Title: A Multicenter, Open Label, Randomized, Comparative Study to Evaluate the Efficacy and Safety of Electric Smart Insulin Pen DIA:CONN P8 in Patients With Type 1, Type 2 or Pancreatogenic Diabetes Mellitus Under Multiple Dose Insulin Therapy
Brief Title: DIA:CONN P8(Smart Insulin Pen) Study in Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G2e Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P8_S301
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Diabetes (Insulin-requiring, Type 1 or Type 2); Pancreatogenic Diabetes Mellitus
Keywords: smart insulin pen; smart insulin pen with dose calculator; insulin dose calculator
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): For the treatment group, education sessions will be conducted during the baseline visit on carb counting and bolus calculator methods, installation, and usage instructions for DIA:CONN P8 and DIA:CONN app, as well as CGM and CGM app. During the 12-week, for basal insulin, the treatment group will input and inject the dosage using the DIA:CONN P8, using only the insulin injection and injection recording functions, same as the blind CGM period. For bolus insulin, when the carbohydrate counting is entered or the type of meal is selected into the DIA:CONN P8 application, the insulin dosage is automatically calculated and set using the entered information and other indicators. Subjects inject the insulin at that calculated dosage using the DIA:CONN P8. Insulin injection dosage, time stamps, and other related details will be recorded into DIA:CONN P8 device and app.
  Interventions: Device: Smart Insulin Pen
- Control Group (Other): The control group will receive education on insulin pen and CGM usage, maintaining their conventional multiple dose insulin therapy while implementing CGM. During the 12-week, the control group will use DIA:CONN P8 to manually input and inject the dosage of both basal and bolus insulin, only using the insulin injection and injection recording functions, same as the blind CGM period. Insulin injection dosage, time stamps, and other related details will be recorded into DIA:CONN P8 device and app.
  Interventions: Device: Injection of bolus insulin via conventional therapy using insulin pen

INTERVENTIONS:
Device: Smart Insulin Pen — During the 12-week, for basal insulin, the treatment group will input and inject the dosage using the DIA:CONN P8, using only the insulin injection and injection recording functions, same as the blind CGM period. For bolus insulin, when the carbohydrate counting is entered or the type of meal is selected into the DIA:CONN P8 application, the insulin dosage is automatically calculated and set using the entered information and other indicators. Subjects inject the insulin at that calculated dosage using the DIA:CONN P8.
  Other Names: DIA:CONN P8
  Arms: Treatment Group
Device: Injection of bolus insulin via conventional therapy using insulin pen — During the 12-week, the control group will use DIA:CONN P8 to manually input and inject the dosage of both basal and bolus insulin, only using the insulin injection and injection recording functions, same as the blind CGM period.
  Arms: Control Group

SUMMARY:
A Multicenter, Open label, Randomized, Comparative Study to Evaluate the Efficacy and Safety of Electric Smart Insulin Pen DIA:CONN P8 in patients with Type 1, Type 2 or Pancreatogenic Diabetes Mellitus under Multiple Dose Insulin Therapy

DETAILED DESCRIPTION:
[Blind CGM Period] All eligible participants who voluntarily provide informed consent to participate in this clinical trial and are determined suitable for trial inclusion/exclusion criteria undergo a blind CGM before the baseline visit (randomization). During this period, every subjects is provided with two DIA:CONN P8 devices for continuous glucose monitoring (CGM), basal insulin, and bolus insulin administration.

Throughout this period, subjects receive training on fundamental insulin pen usage and CGM operation. They use the DIA:CONN P8 specifically for insulin dosage entry and administration, functioning similarly to a conventional insulin pen, only utilizing the injection and injection recording function.

Insulin injection dosages and timing (time stamps) recorded on the DIA:CONN P8 and the participant's blood glucose data logged in the CGM app are collected.

[Application Period] The subject allocated to the intervention or control group through randomization will visit hospital maximun 5 times during the 12-week application period, including the baseline visit, in the following process.

1. Treatment Group: For the treatment group, education sessions will be conducted during the baseline visit on carb counting and bolus calculator methods, installation, and usage instructions for DIA:CONN P8 and DIA:CONN app, as well as CGM and CGM app.
2. Control Group: The control group will receive education on insulin pen and CGM usage, maintaining their conventional multiple dose insulin therapy while implementing CGM.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 19 and 75 years old.
2. Confirmed diagnosis of Type 1 or Type 2 diabetes or post-pancreatectomy(total or partial) diabetes at least 1 year prior to screening.
3. Currently using multiple dose insulin therapy at least 3 months prior to screening, regardless of Continuous Glucose Monitoring(CGM) usage.
4. HbA1c levels between 7.5% and 12.0% at screening.

Exclusion Criteria:

1. Who have administered medications affecting glucose metabolism within 3 months before screening(e.g., corticosteroids, immunosuppressants) (Candidate with stable, ongoing dosage for over 6 months before screening are exempted from this criterion).
2. Diagnosed with clinically significant cardiovascular disease within 6 months prior to screening.
3. Exhibiting an estimated glomerular filtration rate(eGFR)<15 mL/min at the screening.
4. Unable to engage in study education due to severe systemic disorders(e.g., end-stage renal failure requiring dialysis, liver cirrhosis of Child-Pugh Class C or higher, etc)
5. Participants with severe diabetic complications(e.g., diabetic foot, diabetic retinopathy, etc)
6. Pregnant or lactating women

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c(%) at 12 weeks compared to baseline | from baseline to the 12-week time point
  Descriptive statistics (sample size, mean, standard deviation, median, minimum, and maximum) are provided for the change in HbA1c (%) from baseline to the 12-week time point, stratified by group.

CONTACTS AND LOCATIONS:
Overall Officials: TAEMIN LEE, Study Director — G2e Co., Ltd
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No